CLINICAL TRIAL: NCT05159011
Title: Access to Genetic Information Leveraging Innovative Technology
Brief Title: Access to Genetic Information Leveraging Innovative Technology (AGILITY)
Acronym: AGILITY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never enrolled.
Sponsor: RTI International (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 202100637
Record Dates: First submitted 2021-10-27; First posted 2021-12-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Genetic Testing

STUDY DESIGN:
Intervention Model Description: Interventional chat bot
Who Masked: Investigator
Masking Description: Investigator masked from randomization until results analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Virtual Genetic Counseling
- Chatbot (Other): computer program that that uses machine learning to provide tailored counseling to patients
  Interventions: Behavioral: AGILITY (Access to Genetic Information Leveraging Innovative TechnologY)

INTERVENTIONS:
Behavioral: AGILITY (Access to Genetic Information Leveraging Innovative TechnologY) — information about genetic testing through technology
  Other Names: Chatbot
  Arms: Chatbot

SUMMARY:
AGILITY is a type 1 hybrid trial that will test the effectiveness of a chatbot to provide pre-test information about genetic screening for tier 1 conditions. A randomized control trial of 2400 adult participants from diverse primary care clinics at the University of Florida Gainesville to receive virtual information about tier 1 condition genetic testing from a chatbot or traditional genetic counseling. The assessment of the outcome of the trial is to determine whether the chatbot is inferior to genetic counseling. Non-inferiority will be determined based on informed choice to undergo testing (or not). Implementation outcomes of acceptability, feasibility, and appropriateness will be evaluated to inform future potential through interviews with patients, primary care providers and GCs.

DETAILED DESCRIPTION:
AGILITY is a type 1 hybrid trial that will test the effectiveness of a chatbot to provide pre-test information about genetic screening for tier 1 conditions. A randomized control trial of 2400 adult participants from diverse primary care clinics at the University of Florida Gainesville to receive virtual information about tier 1 condition genetic testing from a chatbot or traditional genetic counseling. The assessment of the outcome of the trial is to determine whether the chatbot is inferior to genetic counseling. Non-inferiority will be determined based on informed choice to undergo testing (or not). Implementation outcomes of acceptability, feasibility, and appropriateness will be evaluated to inform future potential through interviews with patients, primary care providers and GCs. This trial will provide evidence of whether chatbots can serve to address a shortage of genetic counselors by extending pre-test education in a population screening environment to alternate sources such as chatbots. Inclusion of an observation arm for individuals with positive family history who then are offered traditional clinical genetic service is a strength of the design that will allow for contrast between populations and service models as well. Inclusion of assessments of feasibility, acceptability, and appropriateness from multiple stakeholders is critical to future study design and implementation potential.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male or Female
* University of Florida Gainesville primary care patients
* Negative family history for hereditary breast and ovarian cancer, and Lynch syndrome and familial hypercholesterolemia

Exclusion Criteria:

* Positive family history of hereditary breast and ovarian cancer, and Lynch syndrome, and familial hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Informed Choice | Immediately after arm completion
  The number of participants that made an informed choice (Multi-dimensional Model of Informed Choice) following a chatbot intervention compared to the number of participants that made an informed choice following genetic counseling. Informed choice is measured using a composite tool that includes understanding of relevant knowledge (1-8 items-higher scores indicate greater knowledge), attitudes toward testing (1-5 items-higher scores represent more positive attitudes), and whether the test decision is congruent with personal values (positive or negative about testing in relation to whether testing was accepted or declined).

SECONDARY OUTCOMES:
Test-related Affect | 3 months
  Compare Test-related affect scale response assessed by the Feelings About Genomic Testing Results Scale (Response ranges 0-12 on the negative emotions subscale, 0-16 on the positive feelings subscale, 0-12 on the uncertainty subscale, and 0-8 on the privacy concerns subscale, all with a higher score indicating greater functional impairment.) between usual care and the intervention group at 3 months.
Test-related Affect | 6 months
  ompare Test-related affect scale response assessed by the Feelings About Genomic Testing Results Scale (Response ranges 0-12 on the negative emotions subscale, 0-16 on the positive feelings subscale, 0-12 on the uncertainty subscale, and 0-8 on the privacy concerns subscale, all with a higher score indicating greater functional impairment.) between usual care and the intervention group at 6 months.
Decisional Conflict | 3 months
  Compare Decisional conflict assessed by the Ottawa Decisional Conflict Scale (Response range 1-10 higher scores denote greater decisional conflict) between usual care and the intervention group at 3 months.
Decisional Conflict | 6 months
  Compare Decisional conflict assessed by the Ottawa Decisional Conflict Scale (Response range 1-10 higher scores denote greater decisional conflict) between usual care and the intervention group at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Biesecker, PhD, Principal Investigator — RTI International; Alexander S Parker, PhD, Principal Investigator — University of Florida

REFERENCES:
- [Background] Turbitt E, Chrysostomou PP, Peay HL, Heidlebaugh AR, Nelson LM, Biesecker BB. A randomized controlled study of a consent intervention for participating in an NIH genome sequencing study. Eur J Hum Genet. 2018 May;26(5):622-630. doi: 10.1038/s41431-018-0105-7. Epub 2018 Feb 16. PMID 29453419
- [Background] Lewis MA, Paquin RS, Roche MI, Furberg RD, Rini C, Berg JS, Powell CM, Bailey DB Jr. Supporting Parental Decisions About Genomic Sequencing for Newborn Screening: The NC NEXUS Decision Aid. Pediatrics. 2016 Jan;137 Suppl 1(Suppl 1):S16-23. doi: 10.1542/peds.2015-3731E. PMID 26729698
- [Background] Dormandy E, Hooper R, Michie S, Marteau TM. Informed choice to undergo prenatal screening: a comparison of two hospitals conducting testing either as part of a routine visit or requiring a separate visit. J Med Screen. 2002;9(3):109-14. doi: 10.1136/jms.9.3.109. PMID 12370321
- [Background] Li M, Bennette CS, Amendola LM, Ragan Hart M, Heagerty P, Comstock B, Tarczy-Hornoch P, Fullerton SM, Regier DA, Burke W, Trinidad SB, Jarvik GP, Veenstra DL, Patrick DL. The Feelings About genomiC Testing Results (FACToR) Questionnaire: Development and Preliminary Validation. J Genet Couns. 2019 Apr;28(2):477-490. doi: 10.1007/s10897-018-0286-9. Epub 2018 Dec 14. PMID 30964586
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Ames AG, Jaques A, Ukoumunne OC, Archibald AD, Duncan RE, Emery J, Metcalfe SA. Development of a fragile X syndrome (FXS) knowledge scale: towards a modified multidimensional measure of informed choice for FXS population carrier screening. Health Expect. 2015 Feb;18(1):69-80. doi: 10.1111/hex.12009. Epub 2012 Oct 15. PMID 23067225
- [Background] Jaques AM, Sheffield LJ, Halliday JL. Informed choice in women attending private clinics to undergo first-trimester screening for Down syndrome. Prenat Diagn. 2005 Aug;25(8):656-64. doi: 10.1002/pd.1218. PMID 16049990